CLINICAL TRIAL: NCT03838094
Title: Clinical and Radiographic Evaluation of MTA Versus Biodentine as Pulpotomy Agents in Immature First Permanent Molars: A Randomized Clinical Trial
Brief Title: Evaluation of MTA Versus Biodentine as Pulpotomy Agents in Immature First Permanent Molars
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gihan M Abuelniel ,PhD (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Gihan M Abuelniel ,PhD, Associate Professor of Pediatric Dentistry, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19119
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Carious Exposure of Pulp
Keywords: pulp exposure; vital immature; MTA; Biodentine
MeSH Terms: interventions — tricalcium silicate; Pemetrexed; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTA Group (Active Comparator): pulpotomy technique using fast-setting mineral trioxide aggregate (MTA) to be considered the control group for vital pulp therapy and was placed over the amputated pulps for 18 months. This group will be compared with the Biodentine group as the intervention group
  Interventions: Biological: MTA
- Biodentine group (Experimental): 3 mm- thick Biodentine covered radicular pulp to allow pulp regeneration
  Interventions: Biological: Biodentine

INTERVENTIONS:
Biological: Biodentine — it is a dentin substitute, a new biologically active material facilitates its penetration through opened dentinal tubules to crystallize interlocking with dentin and provide mechanical properties.
  Other Names: Calcium silicate-based biomaterial
  Arms: Biodentine group
Biological: MTA — MTA is a powder that consists of fine hydrophilic particles that set in the presence of moisture. MTA consists of tricalcium silicate, tricalcium aluminate, tricalcium oxide and silicate oxide. MTA was considered a remarkable biocompatible material with various clinical applications that include surgical and non-surgical applications such as pulp capping
  Other Names: mineral trioxide aggregate
  Arms: MTA Group

SUMMARY:
Aim of the study: To compare the clinical and radiographic outcomes of mineral trioxide aggregate (MTA) and Biodentine as vital pulp therapy materials (pulpotomy) of cariously exposed vital immature mandibular first permanent molars.

Materials and Methods: sixty immature first mandibular permanent molars cariously exposed with symptomatic /asymptomatic pulpitis were included in the study according to inclusion criteria and were equally divided in two groups. Following split-mouth design molars were randomly assigned to either a control group (MTA 30 molars) or a test group (Biodentine 30 molars). After conducting pulpotomy and covering pulp stumps with the MTA and Biodentine, treated molars received permanent restorations. Blinded clinical and radiographic evaluations were performed at different time intervals (base line immediate postoperative, 6, 12 and 18 months) according to clinical and radiographic criteria of success. Data were recorded and analysed.

DETAILED DESCRIPTION:
Diagnosis:

1. Full history data will be collected, including personal, medical and previous dental data
2. Clinical examination using mirror and probe to assess the inclusion criteria.
3. Radiographic examination using preoperative digital periapical radiograph to assess the inclusion criteria.
4. Preoperative photograph will be taken.

Operative procedure:

Experimental group:

1. Injection of local anesthesia and rubber dam isolation.
2. caries and roof of the pulp chamber will be removed by a fissure diamond bur (Diatech, Heerbrug, Switzerland) and high-speed handpiece with coolant.
3. The pulps will be amputated to the orifice level using a long-shank diamond round bur.
4. Haemostasis will be achieved by gentle placement of a saline-moistened cotton pellet over amputated pulps for 5-10 min.
5. Calcium silicate-based BiodentineTM (Septodont Ltd., Saint Maur des Fausse´s, France) will be mixed according to the manufacturer's instructions, radicular pulp will be covered by the material using a wet cotton pellet.
6. A self-cure glass ionomer (GC; GC Corporation, Tokyo, Japan) will be placed over the pulpotomy agent as a final restoration.
7. Immediate post-operative radiograph and photograph will be taken.

Control group:

The same procedures will be carried out as the experimental group, but the pulp stumps will be covered with fast-setting mineral trioxide aggregate (MTA) ENDOCEM MTA (Maruchi, Wonju, Korea) and will be prepared according to the manufacturer's instructions. A 3-mm-thick layer of MTA will be placed over the amputated pulps and will be gently adapted to the dentinal walls using a wet cotton pellet. A self-cure glass ionomer (GC; GC Corporation, Tokyo, Japan) will be placed over the pulpotomy agent as a final restoration.

Postoperative care:

Instructions to avoid lip and cheek biting in addition to oral hygiene measures.

Follow up:

Assess the outcomes clinically and radiographically at (baseline, 6, 12 and 18 months).

ELIGIBILITY:
Inclusion Criteria:

* Bilaterally Symptomatic ⁄ asymptomatic vital immature mandibular first permanent molars (with clinical carious exposure of the pulp and presence of bleeding upon exposure)

  * Patients with an age range from 7-8 years.
  * Absence of sinus tract, soft tissue swelling.

Exclusion Criteria:

* • Molars were excluded if non-restorable.

  * excessive mobility (more than 1 mm horizontally).
  * Radiographic evidence of peri- and ⁄or inter-radicular lesions, internal⁄ external root resorption, pulp⁄ canal calcifications.

Ages: 7 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
pain, sensitivity to percussion⁄ palpation | 18 months
  by asking the patient( binary measure)Yes or No, where Yes indicates presence of pain that shows clinical failure
Swelling or sinus tract | 18 months
  by visual examination( Binary measure) (Yes or No) where No indicates success of the treatment
tooth mobility | 18 months
  by back of the mirror( Binary measure) (Yes or No) where No mobility indicates success of the treatment

SECONDARY OUTCOMES:
root formation/development stage | 18 months
  by radiographic parallel technique to measure the maturity scores used during the radiographic assessment of root development are F, G and H (where F is the worse and H is the best stage)
Crown: Root ratio | 18 months
  by radiographic parallel technique ( the ratio 2:1 or more than 2:1) the ratio more than 2:1 is the best
Apical closure | 18 months
  by radiographic parallel technique( the apex is blunder apex ,partially open, or constricted) blunder apex is the worse and constricted apex is the best.
presence of radiolucency | 18 month
  by radiographic parallel technique( binary measure)( yes or No) if radiolucency is detected this indicates failure of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gihan M Abuelniel, PhD, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No
only final results

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT03838094/Prot_SAP_000.pdf